CLINICAL TRIAL: NCT00368537
Title: A Multicenter, Randomized, Open-Label Comparison of the Safety And Efficacy of Tigecycline With That of Ampicillin-Sulbactam or Amoxicillin-Clavulanate to Treat Complicated Skin And Skin Structure Infections
Brief Title: Study Comparing the Safety and Efficacy of Tigecycline With Ampicillin-Sulbactam or Amoxicillin-Clavulanate to Treat Skin Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3074A1-900
Record Dates: First submitted 2006-08-21; First posted 2006-08-24 (Estimated); Results first posted 2012-08-09 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Skin Diseases, Bacterial
Keywords: skin infection; antibiotics
MeSH Terms: conditions — Skin Diseases, Bacterial; Cellulitis | interventions — Tigecycline; sultamicillin

ARMS (2):
- 1 (Active Comparator): Arm 1: Tigecycline
  Interventions: Drug: Tigecycline
- 2 (Active Comparator): Arm 2: Ampicillin-Sulbactam or Amoxicillin-Clavulanate plus or minus a glycopeptide
  Interventions: Drug: ampicillin-sulbactam

INTERVENTIONS:
Drug: Tigecycline — Treatment A: Tigecycline every 12 hours intravenous (IV) (an initial dose of 100 mg followed by 50 mg every 12 hours)
  Arms: 1
Drug: ampicillin-sulbactam — Ampicillin-sulbactam: 1.5 g (1 g ampicillin plus 0.5 g sulbactam) to 3 g (3 g ampicillin plus 1 g sulbactam) intravenous (IV) every 6 hrs or Amoxicillin-clavulanate: 1.2 g (1000 mg amoxicillin plus 200 mg clavulanate) IV every 6 to 8 hrs.
  A glycopeptide antibiotic (either vancomycin 1 g IV every 12 hrs or teicoplanin IV loading dose of 400 mg the first day followed by a maintenance dose of 200 mg daily) may be added to the aminopenicillin/betalactamase inhibitor regimen if infection with methicillin-resistant staphylococcus aureus (MRSA) is suspected or confirmed within the first 72 hrs of enrollment. If culture results fail to show a resistant organism, use of the glycopeptide may be discontinued.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the safety and efficacy of the antibiotic tigecycline with other antibiotics, ampicillin-sulbactam, and amoxicillin-clavulanate in the treatment of a complicated skin and/or skin structure infection (cSSSI).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of complicated skin or skin structure infection
* Male or female, 18 years or older
* Need for intravenous treatment for 4 to 14 days

Exclusion Criteria:

* Skin infection that can be treated by surgery & wound care alone
* Diabetic foot ulcers or bedsores where the infection is present longer than 1 week
* Poor circulation such that amputation of the infected site is likely within a month Other exclusions apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Hong Kong: medinfo@wyeth.com; Trial Manager, Principal Investigator — For South Africa: ZAFinfo@wyeth.com; Trial Manager, Principal Investigator — For Taiwan: medinfo@wyeth.com
Locations (52):
- United States (30):
  - Scottsdale, Arizona
  - Jonesboro, Arkansas
  - Chula Vista, California
  - Mission Viejo, California
  - National City, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Vero Beach, Florida
  - Fort Eisenhower, Georgia
  - Idaho Falls, Idaho
  - Decatur, Illinois
  - Naperville, Illinois
  - Springfield, Illinois
  - Topeka, Kansas
  - Cambridge, Massachusetts
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Lincoln, Nebraska
  - Hackensack, New Jersey
  - Neptune City, New Jersey
  - Buffalo, New York
  - Elmira, New York
  - New Hyde Park, New York
  - Columbus, Ohio
  - Lima, Ohio
  - Lansdale, Pennsylvania
  - Philadelphia, Pennsylvania
  - Fort Worth, Texas
  - Houston, Texas
- Canada (7):
  - Winnipeg, Manitoba
  - Chicoutimi, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
  - Trois-Rivières, Quebec
  - Saskatoon, Saskatchewan
- Hong Kong, Hong Kong
- Ramat Gan, Israel
- Beirut, Lebanon
- Pulau Pinang, Malaysia
- Manila, Philippines
- Singapore, Singapore
- South Africa (4):
  - Cape Town
  - Gauteng
  - KZ-Natal
  - Mpumalanga
- South Korea (3):
  - Daejeon
  - Incheon
  - Seoul
- Taipei, Taiwan
- Bangkok, Thailand

REFERENCES:
- [Derived] Matthews P, Alpert M, Rahav G, Rill D, Zito E, Gardiner D, Pedersen R, Babinchak T, McGovern PC; Tigecycline 900 cSSSI Study Group. A randomized trial of tigecycline versus ampicillin-sulbactam or amoxicillin-clavulanate for the treatment of complicated skin and skin structure infections. BMC Infect Dis. 2012 Nov 12;12:297. doi: 10.1186/1471-2334-12-297. PMID 23145952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited worldwide from September 2006 to August 2008.
Pre-assignment Details: Patients were screened according to the inclusion/exclusion criteria. Once informed consent was obtained, the patient was enrolled into the study and assigned a randomization number and a treatment regimen.
Groups:
- Tigecycline: Tigecycline every 12 hours IV (an initial dose of 100 mg followed by 50 mg every 12 hours)
- Ampicillin-Sulbactam or Amoxicillin-Clavulanate: Ampicillin-sulbactam 1.5 g (1 g ampicillin plus 0.5 g sulbactam) to 3 g (2 g ampicillin plus 1 g sulbactam) IV every 6 hours or amoxicillin-clavulanate 1.2 g (1000 mg amoxicillin plus 200 mg clavulanate) IV every 6 to 8 hours.
Period: Randomization
Arm/Group | Tigecycline | Ampicillin-Sulbactam or Amoxicillin-Clavulanate
Started | 281 | 269
Completed | 268 | 263
Not Completed | 13 | 6
Not completed — No study drug dosed | 13 | 6
Period: Baseline Participants
Arm/Group | Tigecycline | Ampicillin-Sulbactam or Amoxicillin-Clavulanate
Started | 268 | 263
Completed | 244 | 239
Not Completed | 24 | 24
Not completed — Lost to Follow-up | 16 | 17
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Death | 1 | 2
Not completed — No susceptibility | 1 | 0
Not completed — Patient uncompliant | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tigecycline | Ampicillin-Sulbactam or Amoxicillin-Clavulanate | Total
Number analyzed (Participants) | 268 | 263 | 531
Age Continuous [Mean (Standard Deviation); unit: years] | 51.10 (16.11) | 51.54 (16.90) | 51.32 (16.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 94 | 199
  Male | 163 | 169 | 332

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinically Evaluable (CE) Patients With Clinical Response of Cure at the Test-of-cure (TOC) Visit
Description: Investigator assigned clinical response of cure of the cSSSI defined as: resolution of all clinical signs and symptoms of infection (healing of chronic underlying skin ulcer not required) or improvement of signs or symptoms of the infection to such an extent that no further antibacterial therapy was necessary. CE population were those who completed TOC assessment of cure or failure (but not indeterminate) or, in case of premature discontinuation due to lack of efficacy, had completed end of treatment assessment such that assessment of clinical response could be made.
Time Frame: up to 6 weeks
Population: Clinically Evaluable (CE): Patients with cSSSI, no Pseudomonas aeruginosa as sole baseline isolate, met major inclusion/exclusion criteria, ≤24 hrs antibiotics pre-baseline, had ≥4 days of study drug, compliant with therapy. Excludes indeterminates.
Measure: Number; unit: participants
Arm/Group | Tigecycline | Ampicillin-Sulbactam or Amoxicillin-Clavulanate
Number analyzed (Participants) | 209 | 196
participants | 162 | 152
Statistical Analysis 1: Comparison: Tigecycline vs Ampicillin-Sulbactam or Amoxicillin-Clavulanate; Test type: Non-Inferiority or Equivalence — A 2-sided 95% CI (corrected for continuity) was calculated for the true difference between the cure rates. Non-inferiority will be concluded if the lower limit of the 2-sided CI is greater than -15%; Risk Difference (RD) = 0.0, 95% CI [-8.7 to 8.6] — Confidence interval calculated using asymptotic method corrected for continuity. Difference= Tigecycline minus Ampicillin-Sulbactam or Amoxicillin-Clavulanate

2. Secondary Outcome: Number of Microbiologically Evaluable Patients With Clinical Response of Cure at the Test-of-cure (TOC) Visit
Description: Investigator assigned clinical response of cure of the cSSSI defined as: resolution of all clinical signs and symptoms of infection (healing of chronic underlying skin ulcer not required) or improvement of signs or symptoms of the infection to such an extent that no further antibacterial therapy was necessary. ME population were subjects who were CE and had baseline culture with at least 1 identified isolate that was susceptible to study drug and comparator. TOC performed 8-50 days after last dose of study drug.
Time Frame: up to 6 weeks
Population: Microbiologically Evaluable patients:Clinically Evaluable (CE) patients who had baseline culture with ≥1 identified pathogen susceptible to both study drugs (ie, the pathogen is susceptible to tigecycline and comparator). Excludes indeterminates.
Measure: Number; unit: participants
Arm/Group | Tigecycline | Ampicillin-Sulbactam or Amoxicillin-Clavulanate
Number analyzed (Participants) | 120 | 99
participants | 96 | 77
Statistical Analysis 1: Comparison: Tigecycline vs Ampicillin-Sulbactam or Amoxicillin-Clavulanate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 2.2, 95% CI [-9.6 to 14.0] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Microbiologically Evaluable Patients by Microbiologic Response at Test-of-Cure (TOC) Visit
Description: Microbiological response assessed at patient level. Eradication=baseline isolate not present in repeat culture from the original infection site; Presumed Eradication=clinical response of cure precluded the availability of a specimen for culture; Persistence=baseline isolate present in repeat culture from the original infection site; Presumed Persistence=culture data not available for patients with a clinical response of failure; Superinfection=culture from the primary infection site had new pathogen not identified as a baseline isolate and clinical response was failure.
Time Frame: up to 6 weeks
Population: Microbiologically Evaluable patients:CE patients who had baseline culture with ≥1 identified pathogen susceptible to both study drugs (ie, the pathogen is susceptible to tigecycline and comparator). TOC performed 8-50 days after last dose of study drug.
Measure: Number; unit: participants
Arm/Group | Tigecycline | Ampicillin-Sulbactam or Amoxicillin-Clavulanate
Number analyzed (Participants) | 120 | 99
participants
  Eradication + presumed eradication | 95 | 76
  Persistence + Presumed persistence | 25 | 23
  Superinfection | 2 | 1
Statistical Analysis 1: Comparison: Tigecycline vs Ampicillin-Sulbactam or Amoxicillin-Clavulanate; Group comparison of eradication + presumed eradication; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 2.4, 95% CI [-9.6 to 14.4] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Minimum Inhibitory Concentration (MIC) 50 and 90 by Baseline Isolate
Description: In vitro activity of the study drugs against a range of pathogenic bacteria that cause complicated skin and skin structure infection (cSSSI) were analyzed using MIC. MIC 50 and MIC 90 are the lowest concentrations of a drug that inhibit the growth of 50% and 90% of a microorganism, respectively. TOC performed 8-50 days after last dose of study drug.
Time Frame: up to 6 weeks
Population: m-mITT: Patients with ≥1 dose of study drug, had cSSSI and baseline isolate from infection site / blood. MIC reported for isolates present in ≥10 m-mITT patients. In the categories below "n" is the actual number of isolates used to caluculate the MIC 50 and MIC 90.
Measure: Number; unit: mcg/mL
Arm/Group | Tigecycline | Ampicillin-Sulbactam or Amoxicillin-Clavulanate
Number analyzed (Participants) | 120 | 99
mcg/mL
  Enterococcus Faecalis MIC50 (n=20,20) | 0.12 | 1.00
  Enterococcus Faecalis MIC90 (n=20,20) | 0.25 | 1.00
  Escherichia Coli MIC50 (n=29,29) | 0.25 | 8.00
  Escherichia Coli MIC90 (n=29,29) | 0.50 | 32.00
  Klebsiella Pneumoniae MIC50 (n=13,13) | 0.50 | 2.00
  Klebsiella Pneumoniae MIC90 (n=13,13) | 2.00 | 8.00
  Staphylococcus Aureus MIC50 (n=176,176) | 0.12 | 2.00
  Staphylococcus Aureus MIC90 (n=176,176) | 0.25 | 8.00
  Streptococcus Agalactiae MIC50 (n=18,18) | 0.03 | 0.12
  Streptococcus Agalactiae MIC90 (n=18,18) | 0.06 | 0.12
  Streptococcus Pyogenes MIC50 (n=18,18) | 0.03 | 0.06
  Streptococcus Pyogenes MIC90 (n=18,18) | 0.06 | 0.06

5. Secondary Outcome: Inpatient Healthcare Resource Utilization on or Before Test-of-Cure - Number of Patients
Description: Healthcare resource utilization assessment included intensive care unit (ICU) and non-ICU inpatient hospitalization. TOC performed 8-50 days after last dose of study drug.
Time Frame: up to 6 weeks
Population: All patients who received at least 1 dose of study article.
Measure: Number; unit: participants
Arm/Group | Tigecycline | Ampicillin-Sulbactam or Amoxicillin-Clavulanate
Number analyzed (Participants) | 268 | 263
participants
  Intensive care unit | 6 | 9
  Non-ICU inpatient hospitalization | 268 | 263
Statistical Analysis 1: Comparison: Tigecycline vs Ampicillin-Sulbactam or Amoxicillin-Clavulanate; Intensive care unit; Test type: Superiority or Other; p = 0.444, Fisher Exact; 2-sided; Risk Difference (RD) = -1.2, 95% CI [-4.4 to 2.0]

ADVERSE EVENTS:
Description: This data represents the number of times a given adverse event was reported. The given participant may have experienced more than one adverse event. We are looking at the frequency of adverse events based on event and not by participant.
Arm/Group | Tigecycline | Ampicillin-Sulbactam or Amoxicillin-Clavulanate
Serious Adverse Events (participants affected / at risk) | 38/268 | 29/263
Other Adverse Events (participants affected / at risk) | 396/268 | 241/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tigecycline (N=268) | Ampicillin-Sulbactam or Amoxicillin-Clavulanate (N=263)
Cellulitis (General disorders) | 7 | 6
Infection (General disorders) | 6 | 1
Abscess (General disorders) | 1 | 2
Chest pain (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Carcinoma (General disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Generalized edema (General disorders) | 0 | 1
Overdose (General disorders) | 1 | 0
Retroperitoneal hemorrhage (General disorders) | 1 | 0
Sepsis (General disorders) | 1 | 0
Septic shock (General disorders) | 1 | 0
Traumatic hematoma (General disorders) | 1 | 0
Heart arrest (Cardiac disorders) | 3 | 2
Pulmonary embolus (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Myocardial infarct (Cardiac disorders) | 1 | 0
Occlusion (Vascular disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Cholecystitis (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Esophageal hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hepatic failure (Gastrointestinal disorders) | 0 | 1
Liver function tests abnormal (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Stomach ulcer (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Lung edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Carcinoma of lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute kidney failure (Renal and urinary disorders) | 3 | 1
Kidney failure (Renal and urinary disorders) | 0 | 1
Kidney function abnormal (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Healing abnormal (Metabolism and nutrition disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Herpes simplex (Skin and subcutaneous tissue disorders) | 1 | 0
Necrotising fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
International normalized ratio increased (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tigecycline (N=268) | Ampicillin-Sulbactam or Amoxicillin-Clavulanate (N=263)
Nausea (Gastrointestinal disorders) | 117 | 44
Vomiting (Gastrointestinal disorders) | 64 | 14
Diarrhea (Gastrointestinal disorders) | 38 | 14
Constipation (Gastrointestinal disorders) | 17 | 22
Dyspepsia (Gastrointestinal disorders) | 17 | 7
Headache (General disorders) | 20 | 22
Pain (General disorders) | 15 | 18
Abdominal pain (General disorders) | 17 | 7
Fever (General disorders) | 9 | 6
Chest pain (General disorders) | 5 | 8
Insomnia (Nervous system disorders) | 22 | 17
Anxiety (Nervous system disorders) | 9 | 7
Dizziness (Nervous system disorders) | 9 | 6
Hypokalemia (Metabolism and nutrition disorders) | 6 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 16
Hypertension (Vascular disorders) | 8 | 9
Anemia (Blood and lymphatic system disorders) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.